CLINICAL TRIAL: NCT01495117
Title: Comparison of Chlorhexidine Gluconate and Povidone Iodine as a Preoperative Antisepsis in Clean-contaminated Abdominal Surgery : a Randomized Prospective Trial
Brief Title: Study of Chlorhexidine Gluconate as a Preoperative Antisepsis
Acronym: CHG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seung Duk Lee (Other Government)
Responsible Party: Sponsor-Investigator, Seung Duk Lee, Clinical Fellow, Center for Liver Cancer, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCCCTS-11-563
Record Dates: First submitted 2011-10-14; First posted 2011-12-19 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Surgical Site Infection
Keywords: surgical site infection; chlorhexidine gluconate; povidone iodine
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Povidone Iodine (Active Comparator): 7.5% povidone iodine soaping 10% povidone iodine painting
  Interventions: Drug: Povidone-Iodine
- Chlorhexidine Gluconate (Active Comparator): 4% chlorhexidine gluconate soaping 2% chlorhexidine gluconate painting
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Povidone-Iodine — 7.5% povidone iodine soaping 10% povidone iodine painting
  Other Names: 7.5% POVICLEAN BRUSH (SUNGKWANG PHARM); 10% POVIDONE IODINE SOLUTION (SUNGKWANG PHARM)
  Arms: Povidone Iodine
Drug: Chlorhexidine gluconate — 4% chlorhexidine gluconate soaping 2% chlorhexidine gluconate painting
  Other Names: 4% HEXICLEN BRUSH (SUNGKWANG PHARM); 5% CHLORHEXIDINE GLUCONATE SOLUTION (SUNGKWANG PHARM)
  Arms: Chlorhexidine Gluconate

SUMMARY:
The purpose of this study is to determine which drug (chlorhexidine gluconate vs. povidone iodine) as a preoperative antisepsis in clean-contaminated abdominal surgery (liver, hepatobiliary, small or large bowel, stomach) is effective.

ELIGIBILITY:
Inclusion Criteria:

1. Resection of following organs (clean-contaminated open surgery)

   * Liver, Pancreas, Bile duct, Duodenum
   * Stomach
   * Colon, Small bowel
2. Aged 20 - 85 years old
3. Use Prophylactic antibiotics
4. Use Preoperative bowel preparation
5. Elective operation
6. ASA classification 1-2 ASA I : no known systemic disease ASA II : single systemic disease & mild or well controlled ASA III : multiple systemic diseases or moderately controlled systemic disease ASA IV : poorly controlled systemic diseases
7. adequate organ functions defined as indicated below:

   * WBC 3000 ~ 12 000/mm3
   * > Hb 8.0 g/dl
   * > Plt 100 000/mm3
   * < Cr 1.2 mg/dl

Exclusion Criteria:

1. allergy to chlorhexidine or povidone
2. clean surgery or contaminated surgery
3. patients who cannot be followed up during 1 month
4. patients taking immunosuppressant drugs or chemotherapy agents
5. emergent surgery and reoperation
6. uncontrolled diabetes, BMI > 30 kg/m2
7. vulnerable patients

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with Surgical Site infection within 1month | within 1 month
  Check the surgical site infection (SSI) rate within one month Superficial SSI, Deep SSI, Organ Site SSI decided by physician CDC Definition in 1999 Superficial incisional infection : involving only the skin or subcutaneous tissue of the incision Deep incisional Infection : involving the deep tissues (i.e. fascial and muscle layers) Organ Space Infection : involving any part of the anatomy (i.e. organ/space), other than the incision

SECONDARY OUTCOMES:
Identify the infection source | within 1month
  If SSI occur, we check the infection source including types of bacteriae using culture.
Number of patients with Drug Side effect. | Within 1 month
  We check the side effect of our drugs including chlorhexidine and povidione iodine.
  For example, itching sense, pruritis, ulticaria, redness, anaphylaxis
Number of patients with the postoperative sepsis induced by wound infection | within 1 month
  Definition of Sepsis
  1. Proven infection (by culture, stain) or a clinical syndrome pathognomonic for infection (WBC, imaging finding or petechiae, purpura, or purpura fulminans)
  2. Body temperature (<36 or >38 Celsus Degree)
  3. Heart rate > 90 beats per minute
  4. Respiratory rate > 20 breaths per minute or, on blood gas, a PaCO2 less than 32 mmHg
  5. WBC count <4000 cells/mm3 or >12000 cells/mm3

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Sik Han, Ph.D., Principal Investigator — Liver Cancer Center, National Cancer Center, Republic of Korea
Locations (1):
- National Cancer Center, Republic of Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Park HM, Han SS, Lee EC, Lee SD, Yoon HM, Eom BW, Kim SH, Ryu KW, Park SJ, Kim YW, Park B. Randomized clinical trial of preoperative skin antisepsis with chlorhexidine gluconate or povidone-iodine. Br J Surg. 2017 Jan;104(2):e145-e150. doi: 10.1002/bjs.10395. Epub 2016 Nov 23. PMID 27879993